CLINICAL TRIAL: NCT02579629
Title: Multimodal Post-Cesarean Analgesia With Spinal Morphine and Continuous Wound Infiltration of Ropivacaine Using the OnQ® Elastomeric Pump: A Dose-Ranging Study Using a High-Volume, Low-Dose Protocol
Brief Title: Use of On-Q Pump for Pain Post C-Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, James Dolak, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00073292
Record Dates: First submitted 2015-08-25; First posted 2015-10-19 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Pain
Keywords: Analgesia; Cesarean section; Opiates
MeSH Terms: conditions — Pain; Agnosia | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ropivacaine 0.1% (Active Comparator): Subjects undergoing their first,second or third cesarean sections will receive a bolus dose of 8ml of 0.1% ropivacaine followed by an infusion of 8ml/hr of 0.1% ropivacaine using the On-Q® elastomeric pump for 3 days after the cesarean section.
  Interventions: Drug: Ropivacaine 0.1%; Device: On-Q ® elastomeric pump
- Ropivacaine 0.2% (Experimental): Subjects undergoing their first,second or third cesarean sections will receive a bolus dose of 8ml of 0.2% ropivacaine followed by an infusion of 8ml/hr of 0.2% ropivacaine using the On-Q® elastomeric pump for 3 days after the cesarean section.
  Interventions: Drug: Ropivacaine 0.2%; Device: On-Q ® elastomeric pump
- Normal Saline (Active Comparator): Subjects undergoing their first, second or third cesarean sections will receive a bolus dose of 8ml normal saline followed by an infusion of 8ml/hr of normal saline using the On-Q® elastomeric pump for 3 days after the cesarean section.
  Interventions: Drug: Normal saline; Device: On-Q ® elastomeric pump

INTERVENTIONS:
Drug: Ropivacaine 0.1% — Ropivacaine 0.1% is a local anaesthetic drug and will be administered as a single bolus dose of 8ml of 0.1% ropivacaine followed by an infusion of 8ml/hr of 0.1% ropivacaine using the On-Q® elastomeric pump. The bolus dose of 8ml of 0.1% ropivacaine will be administered via a multiport, silver-impregnated catheter (6-10cm) placed above the rectus muscle parallel to the fascial incision, using a preloaded syringe. The infusion will be delivered by the On-Q® elastomeric pump pre-set to deliver 8ml/hr of 0.1% ropivacaine for 72 hours post-operatively.
  Other Names: Naropin
  Arms: Ropivacaine 0.1%
Drug: Ropivacaine 0.2% — Ropivacaine 0.2% is a local anaesthetic drug and will be administered as a single bolus dose of 8ml of 0.2% ropivacaine followed by an infusion of 8ml/hr of 0.2% ropivacaine using the On-Q® elastomeric pump. The bolus dose of 8ml of 0.2% ropivacaine will be administered via a multiport, silver-impregnated catheter (6-10cm) placed above the rectus muscle parallel to the fascial incision, using a preloaded syringe. The infusion will be delivered by the On-Q® elastomeric pump pre-set to deliver 8ml/hr of 0.2% ropivacaine for 72 hours post-operatively.
  Other Names: Naropin
  Arms: Ropivacaine 0.2%
Drug: Normal saline — Normal saline will be administered as a single bolus dose of 8ml of normal saline followed by an infusion of normal saline using the On-Q® elastomeric pump. The bolus dose of 8ml of normal saline will be administered via a multiport, silver-impregnated catheter (6-10cm) placed above the rectus muscle parallel to the fascial incision, using a preloaded syringe. The infusion will be delivered by the On-Q® elastomeric pump pre-set to deliver 8ml/hr normal saline for 72 hours post-operatively.
  Arms: Normal Saline
Device: On-Q ® elastomeric pump — The On-Q® elastomeric pump automatically and continuously delivers a regulated flow of 0.1% or 0.2% ropivacaine or normal saline locally to the surgical site for 72 hours post-operatively. The infusion will be delivered by pre-setting the On-Q® elastomeric pump to deliver at the rate of 8ml/hr for 72 hours post-operatively.
  Other Names: On-Q PainBuster

SUMMARY:
The main purpose of this study is to examine if pain levels treated with intrathecal (IT) preservative-free morphine (PFM) after a cesarean section improve with the additional use of continuous subfascial wound infiltration with ropivacaine using the OnQ® elastomeric pump system.

DETAILED DESCRIPTION:
The main purpose of this study is to examine if pain levels treated with intrathecal (IT) preservative-free morphine (PFM) after a cesarean section improve with the additional use of continuous subfascial wound infiltration with ropivacaine using the OnQ® elastomeric pump system. As a double-blinded, randomized, placebo controlled study, women undergoing first, second or third cesarean section will be randomly assigned to one of 3 different groups. Group 1 will receive saline, group 2 will be given ropivacaine 0.1%, group 3 will be given ropivacaine 0.2%, all at a rate of 8ml/hr via the OnQ® pump system. Each group will also receive an 8mL bolus of the previously assigned infusate. The investigator will assess pain at rest and with movement at different time periods during the recovery process through 3 months post operatively. The investigator will also assess if the use of this system decreases the need for other pain medications and reduces the potential side-effects of pain treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients at Emory University Hospital Midtown undergoing non-emergent, scheduled or unscheduled first, second or third Cesarean sections
2. Patients who are American Society of Anesthesiology (ASA) Class I-III
3. Patients are at least 34 weeks pregnant
4. Patients to receive spinal anesthesia for their procedure
5. Patients who are 18 years of age or older
6. Patient willing and able to provide written informed consent

Exclusion Criteria:

1. Patients with 3 or more prior Cesarean sections
2. Patients undergoing emergent cesarean section with or without general anesthesia
3. Patients with known allergy to morphine, ketorolac, and/or amide local anesthetics
4. Patients who will not receive spinal anesthesia
5. Patients who are less than 34 weeks pregnant
6. Patients with significant maternal cardiac, liver or renal disease
7. Patients with maternal history of narcotic abuse or dependency
8. Patient with pre-operative fever (>100.4 degrees F)
9. Patients less than 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07; Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Dolak, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between July 2015 and July 2019.
Groups:
- Ropivacaine 0.1%: Subjects undergoing cesarean sections will receive a bolus dose of 8ml of 0.1% ropivacaine followed by an infusion of 8ml/hr of 0.1% ropivacaine using the On-Q® elastomeric pump for 3 days after the cesarean section.
- Ropivacaine 0.2%: Subjects undergoing cesarean sections will receive a bolus dose of 8ml of 0.2% ropivacaine followed by an infusion of 8ml/hr of 0.2% ropivacaine using the On-Q® elastomeric pump for 3 days after the cesarean section.
- Normal Saline: Subjects undergoing cesarean sections will receive a bolus dose of 8ml normal saline followed by an infusion of 8ml/hr of normal saline using the On-Q® elastomeric pump for 3 days after the cesarean section.
Period: Overall Study
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Started | 22 | 20 | 22
Completed | 20 | 19 | 20
Not Completed | 2 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Screen Failure | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Participants that completed the trial were included the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline | Total
Number analyzed (Participants) | 20 | 19 | 20 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (4.7) | 32.1 (5.1) | 31.9 (5.7) | 31.2 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 20 | 59
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 19 | 18 | 19 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 13 | 14 | 42
  White | 1 | 5 | 4 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 20 | 59

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Scores During Cough From Baseline
Description: The intensity of pain during cough will be measured using a visual analogue pain scale (VAPS). Subjects will be instructed to indicate the intensity of the pain by marking on a 100-mm vertical lines with terms describing the extremes of pain intensity. The lines are anchored with "no pain" at the bottom and "worst imaginable pain" at the top. Pain scores range from 0-100, so the change in pain score (post- minus pre-) can theoretically range from -100 to 100. A negative score indicates an improvement in pain. Higher scores indicate higher intensities of pain.
Time Frame: 2 hours post baseline, 6, 12, 24, 48, 72 hours post baseline
Population: The drop of participants at 72 hours reflects patients who were discharged early, prior to the 72 hr Visit. Other missing values occurred when patients could not be located at the scheduled time because they were not in their room.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 20 | 19 | 20
score on a scale
  Change in score at 2-hours post baseline: number analyzed (Participants) | 19 | 19 | 20
  Change in score at 2-hours post baseline | 4 [0 to 15] | 1 [-4.5 to 18.5] | 20.5 [4.75 to 36.25]
  Change in score at 6-hours post baseline: number analyzed (Participants) | 19 | 19 | 20
  Change in score at 6-hours post baseline | 10 [4 to 27] | 3 [-8 to 10] | 10.5 [3.75 to 30.75]
  Change in score at 12-hours post baseline | 14.5 [4 to 26] | 2 [-4 to 13] | 15.5 [9.75 to 41.25]
  Change in score at 24-hours post baseline: number analyzed (Participants) | 20 | 18 | 20
  Change in score at 24-hours post baseline | 20 [1.5 to 45.5] | 27 [0 to 36] | 15.5 [9.75 to 41.25]
  Change in score at 48-hours post baseline | 13 [6.5 to 39.75] | 2 [-2.5 to 26.5] | 15 [-0.5 to 35.75]
  Change in score at 72-hours post baseline: number analyzed (Participants) | 16 | 17 | 16
  Change in score at 72-hours post baseline | 6.5 [-1.5 to 32.25] | 0 [0 to 20] | 3 [-1.5 to 15]

2. Primary Outcome: Change in Pain Scores During 20°Straight Leg Raise
Description: The intensity of pain during 20° straight leg raise will be measured using a visual analogue pain scale (VAPS). Subjects will be instructed to indicate the intensity of the pain by marking on a 100-mm vertical lines with terms describing the extremes of pain intensity. The lines are anchored with "no pain" at the bottom and "worst imaginable pain" at the top. Higher scores indicate higher intensities of pain.
Time Frame: Baseline (At zero time, the time of the first dosing using the On-Q catheter), 2, 6, 12, 24, 48, 72 hours post baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 20 | 19 | 20
score on a scale
  Change in score at 2-hours post baseline: number analyzed (Participants) | 19 | 19 | 20
  Change in score at 2-hours post baseline | 4 [1.5 to 12.5] | 5 [0 to 17.5] | 10.5 [1.75 to 31]
  Change in score at 6-hours post baseline: number analyzed (Participants) | 19 | 19 | 20
  Change in score at 6-hours post baseline | 8 [1 to 18] | 0 [-2 to 6.5] | 5 [0.75 to 19.5]
  Change in score at 12-hours post baseline | -6.5 [-22.5 to 0] | 0 [-2.5 to 1.5] | -6.5 [-28.5 to 0]
  Change in score at 24-hours post baseline: number analyzed (Participants) | 20 | 18 | 20
  Change in score at 24-hours post baseline | 9 [0.75 to 23.75] | 0 [0 to 21.25] | 16 [0.75 to 29]
  Change in score at 48-hours post baseline | 9.5 [0.75 to 21.25] | 3 [0 to 22.5] | 17 [0.75 to 27]
  Change in score at 72-hours post baseline: number analyzed (Participants) | 16 | 17 | 16
  Change in score at 72-hours post baseline | 1 [-3 to 8.25] | 3 [0 to 10] | 2.5 [0 to 12]

3. Primary Outcome: Change in Intensity of Pain: Numerical Pain Scale (NPS) From Baseline
Description: Post-operative pain will be measured using a numerical pain scale (NPS). Subjects will be asked to indicate the level of pain with 0 being no pain and 10 being the worst imaginable pain. Higher scores indicate higher intensities of pain. Participants will report intensity of pain at the week 6 and 3 month time points through a telephone call.
Time Frame: 6 weeks, 3 months
Population: The difference reflects the number of patients who were lost to follow up at 6 weeks and 3 months.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 17 | 19 | 17
units on a scale
  Change at 6 weeks post intervention | 3 [0 to 5] | 2 [0 to 4] | 5 [2.5 to 6.5]
  Change at 3 months post intervention: number analyzed (Participants) | 15 | 18 | 14
  Change at 3 months post intervention | 0 [0 to 3] | 0 [0 to 0] | 0 [0 to 0.75]

4. Primary Outcome: Change in Intensity of Pain: VAPS From Baseline
Description: Incisional pain will be measured using a visual analogue pain scale (VAPS). Subjects will be instructed to indicate the intensity of the pain by marking on a 100-mm vertical lines with terms describing the extremes of pain intensity. The lines are anchored with "no pain" at the bottom and "worst imaginable pain" at the top. Pain scores range from 0-100, so the change in pain score (post- minus pre-) can theoretically range from -100 to 100. A negative score indicates an improvement in pain. Higher scores indicate higher intensities of pain. Participants will report intensity of pain 2hrs post intervention, 6hr, 12hr, 24hr, 48hr, and 72hr post-intervention.
Time Frame: 24 hours post-intervention, 48 hrs, and 72hr post-intervention.
Population: The differences in the number of participants reflect patients who were discharged earlier than 72 hours and patients whose assessments could not be completed because they were not available (out of the room, etc). All 0 values are real reports of "no pain", which was the median score for Outcome 3. None of them represent missing values or NA.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 20 | 19 | 20
units on a scale
  Change in score at 24 hours post intervention | 0 [0 to 5.75] | 0 [0 to 13] | 0 [0 to 44.5]
  Change in score at 48 hours post intervention | 0 [0 to 11.25] | 0 [0 to 13.5] | 0 [0 to 12.28]
  Change in score at 72 hours post intervention | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

5. Primary Outcome: Change in McGill Pain Questionnaire Score From Baseline
Description: Pain with movement will be assessed using the self-report mini-McGill pain questionnaire, consisting of the first 15 questions of the McGill questionnaire, scores 0-3 points for each. It can theoretically range from 0 to 45, with 45 correlating with worse pain.
Time Frame: 2 hours post-intervention, 6 hours, 12 hours, 24 hours, 72 hours, 6 weeks, 3 months post-intervention
Population: The differences in number of participants reflect patients who were discharged earlier than 72 hours and patients whose assessments could not be completed because they were not available (out of the room, etc. )
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 20 | 19 | 20
score on a scale
  2 hrs post Baseline: number analyzed (Participants) | 18 | 19 | 20
  2 hrs post Baseline | 1.5 [0 to 4] | 2 [0 to 3.5] | 2 [1 to 3.5]
  6 hrs post Baseline: number analyzed (Participants) | 19 | 19 | 20
  6 hrs post Baseline | 2 [1 to 4.5] | 2 [1 to 2.5] | 2 [0 to 4.25]
  12 hrs post Baseline: number analyzed (Participants) | 19 | 19 | 19
  12 hrs post Baseline | 1 [0 to 3] | 1 [0 to 2] | 2 [1 to 3.5]
  24 hrs post Baseline: number analyzed (Participants) | 20 | 17 | 19
  24 hrs post Baseline | 1.5 [1 to 5.25] | 3 [1 to 5] | 2 [1 to 5]
  48 hrs post Baseline: number analyzed (Participants) | 20 | 19 | 18
  48 hrs post Baseline | 2.5 [1 to 4.25] | 3 [0 to 6] | 2 [1 to 3]
  72 hrs post Baseline: number analyzed (Participants) | 16 | 15 | 15
  72 hrs post Baseline | 2 [1 to 3] | 3 [0 to 4.5] | 1 [0 to 2.5]
  6 weeks post Baseline: number analyzed (Participants) | 17 | 19 | 17
  6 weeks post Baseline | 0 [0 to 1] | 0 [0 to 1.5] | 0 [0 to 1]
  3 months post Baseline: number analyzed (Participants) | 15 | 18 | 14
  3 months post Baseline | 0 [0 to 1] | 0 [0 to 0] | 0 [0 to 1]

6. Primary Outcome: Change in Pain Scores at Rest From Baseline
Description: The intensity of pain at rest will be measured using a visual analogue pain scale (VAPS). Subjects will be instructed to indicate the intensity of the pain by marking on a 100-mm vertical lines with terms describing the extremes of pain intensity. The lines are anchored with "no pain" at the bottom and "worst imaginable pain" at the top. Higher scores indicate higher intensities of pain.
Time Frame: 2 hours post-intervention, 6 hours, 12 hours, 24 hours, 48 hous, 72 hours post baseline
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 20 | 19 | 20
score on a scale
  Change in score at 2-hours post baseline: number analyzed (Participants) | 19 | 19 | 20
  Change in score at 2-hours post baseline | 5 [0 to 23.5] | 0 [-4.5 to 9] | 7 [0 to 27.75]
  Change in score at 6-hours post baseline: number analyzed (Participants) | 19 | 19 | 20
  Change in score at 6-hours post baseline | 3 [0 to 17] | 0 [-7 to 4] | 5.5 [0 to 15.5]
  Change in score at 12-hours post baseline | 5 [0 to 19.25] | 0 [-7.5 to 3.5] | 1.5 [0 to 12.5]
  Change in score at 24-hours post baseline: number analyzed (Participants) | 20 | 18 | 20
  Change in score at 24-hours post baseline | 8 [0 to 32.75] | 5.5 [-0.75 to 16.75] | 4.5 [-3.25 to 17.75]
  Change in score at 48-hours post baseline | 4.5 [0 to 15.75] | 3 [-4 to 13.5] | 2.5 [-5.5 to 22.5]
  Change in score at 72-hours post baseline: number analyzed (Participants) | 15 | 17 | 16
  Change in score at 72-hours post baseline | 0 [0 to 4] | 0 [0 to 7] | 2 [-6.25 to 13.5]

7. Secondary Outcome: Change in Time From Baseline to First Dose of Rescue Medications
Description: The time to dosing with the first rescue medications like, non-steroidal anti-inflammatory drugs and morphine, for breakthrough pain will be noted. A shorter time to dosing indicates an increased intensity of pain. It will be recorded in hours post intervention.
Time Frame: Baseline (At zero time, the time of the first dosing using the On-Q catheter), 72 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 20 | 19 | 19
Hours | 9.05 [1.38 to 12.94] | 3.50 [1.05 to 9.75] | 2 [1.38 to 10.6]

8. Secondary Outcome: Breastfeeding Success
Description: Breastfeeding success will be measured using LATCH scores. The LATCH system assigns a numerical score, 0, 1, or 2, to five key components of breastfeeding: "L" is for how well the infant latches onto the breast, "A" is for the amount of audible swallowing noted, "T" is for the mother's nipple type, "C" is for the mother's level of comfort and "H" is for the amount of help the mother needs to hold her infant to the breast. The theoretical range of the Latch score is 0 to 10. Higher scores indicate higher success with breastfeeding.
Time Frame: In the post-anesthesia care unit (up to 2 hours post-operatively), 72 hours post-operatively
Population: Data was not obtained/recorded by nurses during shift and some patients were not available (out of the room, etc).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 7 | 6 | 7
score on a scale
  2 hours post intervention: number analyzed (Participants) | 3 | 4 | 2
  2 hours post intervention | 10 [8.75 to 10] | 6.5 [5 to 7.25] | 6.5 [6.25 to 6.75]
  72 hours post intervention | 10 [8.75 to 10] | 10 [9.25 to 10] | 10 [9.25 to 10]

9. Secondary Outcome: Number of Participants With Catheter or Infiltrate-related Issues at 24, 48 and 72 Hours Post-intervention
Description: The cesarean section incision and the catheter insertion site will be evaluated. Any catheter or infiltrate-related issues like wound infection and seroma formation will be noted. It will be reported as number of issues. Wounds will be assessed for infection or dehiscence. Clean wound lines with no evidence of infection indicate better healing.
Time Frame: 24 hours, 48 hours, 72 hours post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 20 | 19 | 20
Participants
  24 hours post intervention | 0 | 0 | 0
  48 hours post intervention | 0 | 0 | 0
  72 hours post intervention | 0 | 1 | 0

10. Secondary Outcome: Number of Patients With Wound Dysesthesia, Infection, Dehiscence and Keloid Formation at 6 Weeks and 3 Months Post-intervention
Description: At the 6 week and 3-month follow-up phone calls the participant will be asked about the presence of wound dysesthesia (numbness, tingling, burning, pricking, allodynia, or hyperesthesia), occurrence of infection, dehiscence, and keloid formation.
Time Frame: 6 weeks postintervention, 3 months postintervention
Measure: Count of Participants; unit: Participants
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 20 | 19 | 20
Participants
  6 Weeks- Wound Dysesthesia | 2 | 2 | 6
  6 Weeks- Infection | 0 | 0 | 0
  6 Weeks- Dehiscence | 0 | 0 | 0
  6 Weeks- Keloid Formation | 0 | 0 | 0
  3 Months- Wound Dysesthesia | 1 | 2 | 3
  3 Months - Infection | 0 | 0 | 0
  3 Months- Dehiscence | 0 | 0 | 0
  3 Months- Keloid Formation | 0 | 0 | 0

11. Secondary Outcome: Cost Analysis
Description: A cost analysis will occur for the inpatient stay. Costs to be assessed include cost for preparation of the drugs and devices, monitoring/supervision costs based on nursing and physician interventions and cost of days spent in the hospital.
Time Frame: At the time of hospital discharge (average of 3 days)
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 20 | 19 | 20
Dollars | 27.9 (16.6) | 26.8 (18.8) | 31.6 (19.8)

12. Secondary Outcome: Patient Satisfaction at 72 Hours Post Intervention
Description: Patient satisfaction will be assessed by using the visual analog scale (VAS). The visual analog scale (VAS) for satisfaction is a horizontal line 100mm long. At the beginning and the end, there are two descriptors representing extremes of satisfaction. The subjects will be asked to rate their satisfaction by making a vertical mark on the 100mm line, where, 0= least satisfied and 100=most satisfied. Higher scores indicate higher levels of satisfaction.
Time Frame: 72 hours post-operatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 19 | 17 | 20
units on a scale | 60 (40.15) | 61.53 (39.00) | 48.3 (35.43)

13. Secondary Outcome: Dosing Amount of Non-steroidal Anti-inflammatory Drugs
Description: The total dose of non-steroidal anti-inflammatory drugs (NSAIDs) in mg will be recorded for each of the first three post-operative days and after discharge as indicated, along with a cumulative total. Higher doses of NSAIDs usage indicate higher intensities of pain.
Time Frame: 24 post-operatively, 72 hours post-operatively
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 20 | 19 | 19
mg
  24 hours post intervention | 80 (246) | 211 (645) | 379 (899)
  72 hours post intervention | 2040 (799) | 1726 (1075) | 1095 (1228)

14. Secondary Outcome: Amount of Opioid Use
Description: The amount of opioid use will be quantified in terms of morphine equivalents given in mg both by post
  -operative day and with a cumulative total. Higher amounts of opioid use indicates higher degrees of pain.
Time Frame: 24 post-operatively, 72 hours post-operatively
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
Number analyzed (Participants) | 20 | 19 | 20
mg
  24 hours post intervention | 0.35 (1.77) | 6.45 (27.50) | 1.65 (5.28)
  72 hours post intervention | 24.98 (37.81) | 54.28 (164.3) | 31.25 (41.33)

ADVERSE EVENTS:
Time Frame: Adverse Evens were collected during follow up time (Up to 3 months post intervention).
Arm/Group | Ropivacaine 0.1% | Ropivacaine 0.2% | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/20

LIMITATIONS AND CAVEATS:
Research funded internally,no budget for data collection personnel. For LATCH scores, data not obtained by nurses during shift. Early discharge of many patients prior to the 72 hr time point. Significant patient drop out post hospital discharge.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT02579629/Prot_SAP_000.pdf